CLINICAL TRIAL: NCT03159858
Title: Compassionate Use Treatment for a Single Patient With a Custom Made Branched/Fenestrated Endovascular Device for the Treatment of Complex Abdominal Aortic Aneurysm
Status: No longer available | Type: Expanded Access
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01824
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Complex Abdominal Aortic Aneurysm
Keywords: Complex Abdominal Aortic Aneurysm

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Device: Fenerated AAA Endovascular Graft with H&L-B One Shot Introduction System — The Compassionate Use Request is for the use of the Cook Zenith Fenestrated Endovascular Graft (4 branches) for the treatment of a 70-year-old male patient considered unfit for open surgical repair of his 6cm paravisceral abdominal aortic aneurism (AAA).

SUMMARY:
The FENESTRATED AAA ENDOVASCULAR GRAFT WITH THE H&L-B ONE-SHOT™ INTRODUCTION SYSTEM is neither commercially available or available as part of a clinical trial. IRB approval of this protocol was requested so that Cook, Incorporated may apply to the FDA for approval for one-time use of this patient-specific device for compassionate use for patient AO. It is a custom made endovascular device consisting of4 fenestrations for the celiac, SMA (superior mesenteric) and left and right renal arteries.

DETAILED DESCRIPTION:
The Custom Made Branched/Fenestrated Endovascular Device to be used in this treatment plan is not Food and Drug Administration (FDA)-approved, and is approved for use only in a clinical study. However, the FDA has allowed the use of this device for compassionate use.

The devices used are tubular grafts made of polyester fabric sewn to metal stents. The upper part of the grafts includes fenestrations (holes) that allow the grafts to be located above or near major arteries that branch off of the aorta (celiac artery, superior mesenteric artery (SMA), and renal arteries) without blocking blood flow to them. The celiac artery supplies blood to internal organs including the liver and stomach. The SMA supplies blood to internal organs as well, including parts of the large and small intestines. The renal arteries supply blood to the kidneys. Grafts with branches and/or fenestrations are needed when the aneurysm is located near these major arteries. The major arteries that branch off of the aorta (celiac artery, SMA, and renal arteries) may also be treated using stents (small tubular metal structures) to help keep the arteries open and aligned with the graft fenestrations (holes).

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 70 Years to 70 Years | Sex: Male
Age Groups: Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Neal Cayne, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States